CLINICAL TRIAL: NCT06048224
Title: A Randomized Controlled, Double-blind, Phase III, Multicenter Clinical Study of HS628 Versus Actemra® in Combination With Methotrexate as Therapy in Patients With Moderate to Severe Rheumatoid Arthritis
Brief Title: Phase III Clinical Trial Comparing the Safety, Efficacy, and Immunogenicity of Recombinant Anti-interleukin-6 Receptor Humanized Monoclonal Antibody Injection in Combination With Methotrexate and Jamelor ® in the Treatment of Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang Hisun Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS628-III
Record Dates: First submitted 2023-09-06; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Moderate to Severe Active Rheumatoid Arthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS628 (Experimental): Subjects will receive 8mg/kg intravenous(IV) HS628 at Week 0,Week 4, Week 8, Week 12, Week 16, Week 20,Week 24
  Interventions: Drug: HS628+MTX
- Actemra (Active Comparator): Subjects will receive 8mg/kg intravenous(IV) ACTEMRA® at Week 0,Week 4, Week 8, Week 12, Week 16, Week 20,Week 24
  Interventions: Drug: Actemra +MTX

INTERVENTIONS:
Drug: HS628+MTX — Participants will receive HS628 SC injections Q4W along with MTX orally for 24-week
  Arms: HS628
Drug: Actemra +MTX — Participants will receive tocilizumab SC injections Q4W along with MTX orally for 24-week
  Arms: Actemra

SUMMARY:
This is a multi-center, randomized, double-blind, parallel-group study to evaluate the efficacy and safety of intravenous HS628 in combination with MTX versus Actemra in combination with MTX, in participants with moderate to severe active rheumatoid arthritis (RA) who have inadequate response to current MTX therapy. The study comprises a 24-week treatment phase, followed by a 4-week safety observation period.

ELIGIBILITY:
* Inclusion Criteria:

  1. the person who has signed the informed consent and can complete the test according to the program;
  2. age ≥18 years old and ≤75 years old (subject to the date of signing the informed consent), male or female;
  3. weight ≥30kg;
  4. according to the 2010 ACR/EULAR diagnostic criteria, rheumatoid arthritis was diagnosed with the disease duration ≥ 6 months;
  5. swelling and tenderness joint count ≥ 6 (based on 66 joint counts) and tenderness joint count ≥ 6 (based on 68 joint counts) during the screening period, if both swelling and tenderness are present in the same joint, the joint shall be included in both swelling and tenderness joint count (excluding artificial joints);
  6. C-reactive protein (CRP) ≥10mg/L or erythrocyte sedimentation rate (ESR) > 28mm/hr at the screening stage;
  7. patinents who had received DMARD treatment for at least 3 months before screening visit;
  8. Inadequate response to previous or current methotrexate treatment;
  9. patients who received at least 12 weeks of oral methotrexate treatment (≥ 7.5mg/week) and at least 4 weeks of stable oral dose (methotrexate dose 7.5-25mg/week, with critical value) before random administration;
  10. all non-biological agents DMARD except methotrexate should be discontinued for at least 2 weeks before random administration( In addition, leflunomide should be discontinued for ≥8 weeks, and at least 2 weeks before randomized administration if standard coletenide therapy or activated carbon elution has been followed; Discontinuation of sulfasalazine ≥4 weeks; Yunke withdrawal ≥12 weeks）;
  11. Patinents who will receive oral folic acid treatment (at least 5 mg/ week or a dose determined according to local medical practice) or an equivalent drug (a combination of drugs required for MTX treatment) throughout the study, and the dose of folic acid or an equivalent drug was stable for at least 2 weeks prior to random administration.
  12. biologic DMARD should have been discontinued for at least 2 weeks prior to random administration.For example, adamumab, setuzumab, infliximab and golimumab should be discontinued for ≥8 weeks.Etanercept (enley, esipher, and jeanke), Anbainuo should be discontinued for ≥ 4 weeks;Tofetib and baritinib should be discontinued for ≥2 weeks;
  13. any Chinese herbal medicine, proprietary Chinese medicine or natural medicine for the treatment of RA has been discontinued for at least 2 weeks before random administration;
  14. any non-steroidal anti-inflammatory drug must be given at a stable dose for at least 2 weeks prior to random administration;
  15. at the time of screening, if the subject was taking prednisone or a comparable dose of glucocorticoid, the prerandomized stable dose (prednisone dose ≤10mg/ day) was administered for at least 4 weeks;
  16. Non-lactating women and non-pregnant women (negative blood pregnancy test for women of childbearing age; the subject or his or her spouse will use appropriate and effective contraceptive methods, such as abstinence, oral contraceptives, Iuds, or double barrier methods, during the trial period and for 3 months after the end of the last dose.
* Exclusion Criteria:

  1. Subjects have previously received Tocilizumab treatment or are allergic to any component of Tocilizumab (or investigational drug product);
  2. Subjects with long-term bedridden/wheelchair;
  3. Subjects with inflammatory joint disease other than rheumatoid arthritis in their previous or current medical history; or other systemic autoimmune diseases;
  4. Current symptoms of severe, progressive or uncontrolled diseases of renal, hepatic, hematological, gastrointestinal, pulmonary, cardiac, neurological, or cerebral. Concomitant medical conditions that, in the opinion of the investigator, might place the subject at unacceptable risk for participation in this study;
  5. Subjects with history of severe hypersensitivity or anaphylaxis to human, humanized or mouse monoclonal antibodies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 669 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with an ACR20 response | Week 24
  The ACR 20 responses: greater than or equal to 20 percent improvement in TJC and SJC (28 assessed joints), and 20% improvement in 3 of the following 5 criteria, respectively: 1) PtAAP- VAS, 2) PtGADA-VAS, 3) PhGADA-VAS, 4) HAQ-DI, and 5) CRP or ESR

SECONDARY OUTCOMES:
Proportion of patients with an ACR50, 70 response | Week 24
  The ACR50, 70 responses: greater than or equal to 50, 70 percent improvement in TJC and SJC (28 assessed joints), and 50%, 70% improvement in 3 of the following 5 criteria, respectively: 1) PtAAP- VAS, 2) PtGADA-VAS, 3) PhGADA-VAS, 4) HAQ-DI, and 5) CRP or ESR
Proportion of patients with an ACR20, 50, 70 response | Week 12
  The ACR20, 50, 70 responses: greater than or equal to 20, 50 70 percent improvement in TJC and SJC (28 assessed joints), and 20%, 50%, 70% improvement in 3 of the following 5 criteria, respectively: 1) PtAAP- VAS, 2) PtGADA-VAS, 3) PhGADA-VAS, 4) HAQ-DI, and 5) CRP or ESR
Proportion of patients with DAS28 (ESP、CRP) ≤3.2 and <2.6 | Week 12
  The DAS28-ESR（CRP）score is a measure of the patient's disease activity calculated using the tender joint count on 28 joints (TJC28), swollen joint count on 28 joints (SJC28), patient's global assessment (PGA) of disease activity based on visual analog scale (VAS) and the erythrocyte sedimentation rate (C-reactive protein) in millimeter/hour (mm/hr)（mg/L）. VAS assessments involved a 10 cm horizontal scale from 0 (no disease activity) to 10 (maximum disease activity). Total possible score ranged from 0 to 10. Higher scores represent higher disease activity. A negative change from baseline indicates an improvement
Proportion of patients with DAS28 (ESP、CRP) ≤3.2 and <2.6 | Week 24
  The DAS28-ESR（CRP）score is a measure of the patient's disease activity calculated using the tender joint count on 28 joints (TJC28), swollen joint count on 28 joints (SJC28), patient's global assessment (PGA) of disease activity based on visual analog scale (VAS) and the erythrocyte sedimentation rate (C-reactive protein) in millimeter/hour (mm/hr)（mg/L）. VAS assessments involved a 10 cm horizontal scale from 0 (no disease activity) to 10 (maximum disease activity). Total possible score ranged from 0 to 10. Higher scores represent higher disease activity. A negative change from baseline indicates an improvement
Simplified Disease Activity Index (SDAI)Change From Baseline | Week 12、 Week 24
  SDAI is a numerical sum of 5 outcome parameters: TJC and SJC based on a 28-joint assessment, PtGDA and PGDA assessed on 0-10 cm VAS and CRP in mg/dL. Higher positive value indicates greater extent of positive relationship and higher negative value indicates greater extent of negative relationship.
Clinical Disease Activity Index (CDAI)（Change From Baseline） | Week 12、 Week 24
  The CDAI is a numerical sum of 4 outcome parameters: tender joint count (TJC) and swollen joint count (SJC) based on a 28-joint assessment, patient's global assessment of disease activity (PtGDA) and physician global assessment of disease activity (PGDA) assessed on 0-10 centimeters (cm) visual analogue scale (VAS). Higher scores represent greater affectation due to disease activity.
Change From Baseline in TJC and SJC | Week 24
  The number of tender joints (based on 68 joints) and swollen joints (based on 66 joints) were counted at each visit. TJC was determined by identifying the joints that were painful under pressure or to passive motion, A negative change from baseline indicates an improvement.
Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) | Week 24
  HAQ-DI is a participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week.
Change From Baseline in the Short Form 36 (SF-36) Health Survey | Week 24
  The SF-36 Health Survey uses participant-reported symptoms on 8 subscales to assess health-related quality of life (HRQoL). A clinically relevant improvement in the Physical and Mental Component Scores of the SF-36 was defined as a ≥ 5-point increase from Baseline.
Change From Baseline in CRP | Week 12、Week 24
  as stated above
Change From Baseline in ESR | Week 12、Week 24
  as stated above
Change From Baseline in VAS（PtAAP-VAS、PtGADA-VAS、PhGADA-VAS） | Week 12、Week 24
  as stated above

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China